CLINICAL TRIAL: NCT07284641
Title: Hematopoietic Stem Cell Transplantation (HSCT) for Common Variable Immunodeficiency (CVID) and Other Autoimmune Manifestations of Primary Immune Regulatory Disorders (PIRD)
Acronym: CVID/PIRD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25080140
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Common Variable Immunodeficiency (CVID); Primary Immune Regulatory Disorder; Immune Dysregulation; DiGeorge Syndrome; STAT 1 Gain of Function; STAT 3 Gain of Function; Hypomorphic RAG1 Deficiency; CD40 Ligand Deficiency; Mendelian Susceptibility to Mycobacterial Disease; GATA2 Associated Immunodeficiency; CD40 Deficiency; Hypomorphic RAG2 Deficiency; Immune Dysregulation Polyendocrinopathy Enteropathy X-Linked Syndrome; Omenn Syndrome; Chronic Granulomatous Disease
Keywords: HSCT; CVID; PIRD; primary immune regulatory disorder; common variable immunodeficiency; IPEX like syndromes; Immune dysregulation; polyendocrinopathy; enteropathy; X-linked (IPEX syndrome); DiGeorge Syndrome; Combined Immunodeficiency; Chronic Granulomatous Disease; STAT 1 Gain of Function; STAT 3 Gain of Function; Hypomorphic RAG 1 and RAG 2; CD40 or CD40L deficiency; Mendelian Susceptibility to Mycobacterial Disease; GATA2 Associated Immunodeficiency; Inflamed Cartilage Syndrome (MAGIC)
MeSH Terms: conditions — Common Variable Immunodeficiency; DiGeorge Syndrome; Hyper-IgM Immunodeficiency Syndrome; Immune Dysregulation, Polyendocrinopathy, Enteropathy, X-Linked Syndrome; Severe Combined Immunodeficiency; Granulomatous Disease, Chronic; Intestinal Diseases | interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: single center, open label, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hematopoietic stem cell transplant (HSCT) (Other): The participant will receive an allogenic, fully (8 of 8 match) or partially HLA-matched (6-7/8 HLA-matched), stem cell transplant utilizing a conditioning regimen of alemtuzumab/Campath, anti-thymocyte globulin/rabbit ATG, Fludarabine and Melphalan and total body irradiation
  Interventions: Biological: Hematopoietic stem cell transplant (HSCT)

INTERVENTIONS:
Biological: Hematopoietic stem cell transplant (HSCT) — The participant will receive an allogenic, fully (8 of 8 match) or partially HLA-matched (6-7/8 HLA-matched), stem cell transplant utilizing a conditioning regimen of alemtuzumab/Campath, anti-thymocyte globulin/rabbit ATG, Fludarabine and Melphalan and total body irradiation.

SUMMARY:
This is a research protocol that will examine Hematopoietic Stem Cell Transplantation (HSCT) using a reduced conditioning regimen (RIC) with total body Irradiation (TBI) in those diagnosed with Common Variable Immunodeficiency (CVID) and Other Autoimmune Manifestations of Primary Immune Regulatory Disorders (PIRD).

DETAILED DESCRIPTION:
Hematopoietic stem cell transplant (HSCT) with reduced-intensity conditioning has been demonstrated as the best definitive therapy to correct many of these inheritable immune defects (Common Variable Immunodeficiency (CVID) and Other Autoimmune Manifestations of Primary Immune Regulatory Disorders (PIRD). This is a single center, open label, non-randomized, Phase II study in which subjects receive an allogenic, fully (8 of 8 match) or partially Human Leukocyte Antigen (HLA)-matched (6-7/8 HLA-matched), stem cell transplant utilizing a conditioning regimen of alemtuzumab/Campath, anti-thymocyte globulin/rabbit (ATG), Fludarabine and Melphalan and Total Body Irradiation (TBI). Graft sources include bone marrow or mobilized peripheral blood stem cells from either a related or unrelated donor. After stem cell infusion, subjects are followed for 2 years per standard of care practices.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, parent, or legal guardian must have given written informed consent. For pediatric subjects who are developmentally able, assent or affirmation will be obtained.
2. Male or female, 5 through 40 years old, inclusive, at the time of informed consent.
3. Patients must have evidence of common variable immunodeficiency (CVID) or other autoimmune manifestation of a primary immune regulatory disorder (PIRD). Genetic screening is required by a targeting gene panel to determine presence of genetic variations that may lead to inborn errors of immunity.

   Examples of such diseases include, but are not limited to:
   * Common variable immunodeficiency (CVID)
   * Combined Immunodeficiency (CID)
   * Immune dysregulation polyendocrinopathy enteropathy X-linked (IPEX syndrome), IPEX like syndromes
   * Combined immunodeficiency with defects in T-cell-mediated immunity, including Omenn syndrome and DiGeorge Syndrome
   * Chronic Granulomatous Disease (CGD)
   * Signal Transducer and Activator of Transcription (STAT 1) Gain of Function (STAT1 GOF)
   * Signal Transducer and Activator of Transcription (STAT 3) Gain of Function (STAT3 GOF)
   * Hypomorphic Recombination-Activating Genes (RAG) 1 and RAG 2
   * CD40 or CD40L deficiency
   * Mendelian Susceptibility to Mycobacterial Disease
   * GATA-binding factor 2 (GATA2) Associated Immunodeficiency
   * Mouth and Genital Ulcers with Inflamed Cartilage Syndrome (MAGIC)
4. Must have previously failed, due to lack of response or intolerance, mycophenolate mofetil and a B cell-depleting antibody, such as Rituximab
5. Glomerular Filtration Rate (GFR) ≥50 mL/min/1.73 m2
6. Aspartate Aminotransferase (AST) ≤4x upper limit of normal
7. Alanine Aminotransferase (ALT) ≤4x upper limit of normal
8. Direct bilirubin ≤ 2.5 mg/dL
9. Human Immunodeficiency Virus (HIV) negative by serology and PCR
10. Human T-cell Lymphotropic Virus (HTLV) negative by serology
11. Cardiac ejection fraction ≥ 40% or shortening fraction ≥26%
12. Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1) ≥40% predicted for age
13. Peripheral Capillary Oxygen Saturation (SpO2) of >92% at rest on room air
14. Subjects must be a minimum of 8 weeks post-solid organ transplant prior to start of conditioning, if applicable
15. Negative pregnancy test for females >10 years old or who have reached menarche, unless surgically sterilized.
16. All females of childbearing potential and sexually active males must agree to use a FDA approved method of birth control for up to 12 months after stem cell transplant or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause birth defects.
17. Subject and/or parent guardian informed of the potential risks of infertility following stem cell transplant and advised to discuss sperm banking or oocyte harvesting.
18. Transplant endorsement from clinical immunologist

Exclusion Criteria:

1. Allergy to Dimethylsulfoxide (DMSO) or any other ingredient used in the manufacturing of the stem cell product
2. Uncontrolled systemic infection, as determined by the appropriate confirmatory testing e.g. blood cultures, Polymerase chain reaction (PCR) testing, etc.
3. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 4 weeks of stem cell transplant
4. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the subject's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Survival post-HSCT | 2 years post transplant
  review of the existing medical records to check on the participant's survival status

SECONDARY OUTCOMES:
engraftment, based upon chimerism data | 1 month, 2 months, 3 months, 6 months, 12 months, 18 months, 24 months
  review of chimerism test results in the existing medical records to check on degree of donor engraftment measured by the percentage of donor-derived blood cells in the HSCT recipient
Assess myeloid, B and T cell chimerism | up to 2 years post translant
  review test results from medical records to check how donor and recipient cells populate different immune lineages post-transplant
Assess Immunoglobulin A (IgA), Immunoglobulin (IgM), and Immunoglobulin E (IgE) reconstitution | up to 2 years post transplant
  review of the existing medical records to check on the participant's humoral immune recovery.
independence of immunoglobulin replacement (IVIG, IgG) | 1 and 2 year post transplant
  Determine and probability
incidence of acute graft versus host disease (GVHD) | 6 months post transplant
  grades 3-4
chronic graft-versus-host-disease | 1 year post transplant
  grades 3-4

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — UPMC Children's Hospital of Pittsburgh

IPD SHARING:
Plan to Share IPD: No